CLINICAL TRIAL: NCT02127138
Title: A Prospective Multicenter Randomized Trial Assessing the Efficacy and Safety of Active Transfer of Plaque vs. Provisional T Stenting for the Treatment of Unprotected Distal Left Main Bifurcation Lesions
Brief Title: The Study of Active Transfer of Plaque Technique for Unprotected Distal Left Main Bifurcation Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Anzhen Hospital (Other)
Collaborators: Beijing Jishuitan Hospital (Other); Tianjin First Central Hospital (Other); Tianjin Chest Hospital (Other); Taihe Hospital (Other); The Fourth Affiliated Hospital of Harbin Medical University (Other); General Hospital of Ningxia Medical University (Other); Tangshan Worker's Hospital (Other)
Responsible Party: Principal Investigator, Yang Qing, MD, Beijing Anzhen Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ATP 01
Record Dates: First submitted 2014-04-27; First posted 2014-04-30 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Coronary Heart Disease
Keywords: unprotected distal left main bifurcation lesion; Percutaneous coronary intervention; clinical study; Active Transfer of Plaque （ATP）; Provisional T Stenting
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ATP technique (Experimental): This arm plan to enroll 158 subjects，Sirolimus-eluting Drug stent implantation via Active transfer of Plaque technique in the treatment of unprotected distal left main bifurcation lesions.In the ATP technique treatment of bifurcation lesions, by the balloon pre-dilation in the target side branch, the plaque will be actively transferred from side branch to main vessel. Subsequently, the plaque will be fixed by the expansive stent in main vessel. A stent with stent/artery ratio of 1.1:1 is inflated in MV. Rewire to SB is also left at operator's discretion. FKBI or stent in SB is recommended if there is at least one of following: residual stenosis>70%, >type B dissection and TIMI flow<3.
  Interventions: Device: Sirolimus eluting Drug stent
- Provisional T stenting technique (Active Comparator): This arm plan to enroll 158 subjects.Sirolimus-eluting Drug stent implantation via Provisional T Stenting technique in the treatment of unprotected distal left main bifurcation lesions.Provisional T stenting technique is the typic step-T stenting. In brief, two wires are advanced to distal MV and SB. Pre dilation is left at operator's discretion, however, pre dilating SB is not encouraged. Kissing balloon inflation before stenting MV is left at operator's discretion. A stent with stent/artery ratio of 1.1:1 is inflated in MV. Rewire to SB is also left at operator's discretion. FKBI is recommended if there is at least one of following: residual stenosis>70%, >type B dissection and TIMI flow<3.
  Interventions: Device: Sirolimus eluting Drug stent

INTERVENTIONS:
Device: Sirolimus eluting Drug stent — Use the Sirolimus-eluting Drug stents has been approved by the CFDA，But does not allow use taxol-eluting Drug stents and Drug-eluting stent without Polymer.

SUMMARY:
A Prospective Multi-center Randomized Trial Assessing the Efficacy and Safety of Active Transfer of Plaque vs. Provisional T Stenting for the Treatment of Unprotected Distal Left Main Bifurcation Lesions

DETAILED DESCRIPTION:
It is a prospective, multi-center, randomized, open-label, non-inferiority trial. A total of 316 subjects from around 20 selected hospitals will be randomized on a 1:1 basis to either Active transfer of Plaque (ATP) stenting technique or Provisional T stenting technique.

In the ATP treatment of bifurcation lesions, by the balloon pre-dilation in the target side branch, the plaque will be actively transferred from side branch to main vessel. Subsequently, the plaque will be fixed by the expansive stent in main vessel.As to the provisional T treatment, provisional T stenting is the typic step-T stenting. In brief, two wires are advanced to distal MV and SB. Pre dilation is left at operator's discretion, however, pre dilating SB is not encouraged. Kissing balloon inflation before stenting MV is left at operator's discretion. A stent with stent/artery ratio of 1.1:1 is inflated in MV. Rewire to SB is also left at operator's discretion. FKBI is recommended if there is at least one of following: residual stenosis>70%, >type B dissection and TIMI flow<3.

All patients will be followed clinically at 1-, 6- 12- and 24-month after stent implantation. Repeat angiography will be performed in all patients at 13 months after the index procedure.

The primary endpoint of the trial is the rate of TLR at 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be at least ≥18, ≤80 years of age.
* Patient has Stable/unstable angina or NSTEMI
* Patient has STEMI>24-hour from the onset of chest pain to admission.
* LMb (Medina 0,1,1；1,1,1；0,1,0 ；1,1,0).
* Patient is eligible for elective percutaneous coronary intervention (PCI) .
* Patient is an acceptable candidate for coronary artery bypass grafting (CABG).
* Patient (or legal guardian) understands the trial requirements and treatment procedures and provides written informed consent before any trial-specific tests or procedures are performed; patient is willing to comply with all protocol-required follow-up evaluations

Exclusion Criteria:

* Patient with STEMI (within 24-hour from the onset of chest pain to admission).
* Patient has known allergy to the study stent system or protocol-required concomitant medications that cannot be adequately pre-medicated (everolimus, aspirin, contrast media, acrylic acid, Stainless steel).
* Patient has intolerable to dual anti-platelet therapy.
* Patient has any other serious medical illness that may reduce life expectancy to less than 12 months.
* Patient is pregnant or nursing.
* Patient is participating in another clinical trial that has not reached its primary endpoint within 12 months after the index procedure.
* Patient with severe calcified lesions needing rotational atherectomy.
* Left main In Stent Restenosis.
* Investigator consider that patients don't fit to participate in the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2015-05; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Rate of target lesion revascularization (TLR) at 12-month. | 12 months

SECONDARY OUTCOMES:
Rate of target lesion failure(TLF) at 1-, 6-,12- and 24-month after procedure | Up to 2years
Clinically cardiovascular endpoints at 1-, 6- , 12- and 24-month, including all-cause death, MI and any revascularization. | Up to 2 years
Stent thrombosis which is defined according to Academic Research Consortium (ARC) definition, including definite, probable and possible stent thrombosis. | Up to 2 years
Classification score of Canadian Cardiovascular Society (CCS) angina or Braunwald class. | Up to 2 years
The net gain of lumen diameter; in-segment late loss (LL) and ISR of main vessel and side branch at 13-month. | 13 months

OTHER OUTCOMES:
The release of procedure-related biomarker | baseline
Consumption of devices for surgery procedure | baseline
Amount of contrast agent | baseline
Procedure time | baseline
X-ray exposure time | baseline
X-ray dose | baseline
DAP-total, DAP-record, DAP-fluoro | baseline
contrast induced acute kidney injury (CIAKI) | 3 days after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, MD, PhD, Principal Investigator — Beijing Anzhen Hospital
Locations (1):
- Beijing Anzhen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided